CLINICAL TRIAL: NCT04572048
Title: Longitudinal One Year Vs Single Day NRP Training: a Randomized Controlled Trial.
Brief Title: Longitudinal One Year Vs Single Day NRP Training.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Moussa (Other)
Responsible Party: Sponsor-Investigator, Ahmed Moussa, Principal Investigator, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MP-21-2020-2444
Record Dates: First submitted 2020-09-03; First posted 2020-10-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Nurse Training in Neonatal Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-day NRP training (Other): This group will follow the single-day NRP training course that is currently the standard. It usually takes 8 hours to complete this training course and the nurses are released from their clinical duty to attend the training course.
  Interventions: Other: Single-day NRP Training
- Longitudinal one year NRP Training (Experimental): This group will follow the longitudinal NRP training course. The longitudinal NRP training course will consist of nine 30-minute modules that will be taught every 6-8 weeks over a period of one year. The nurses will attend the different modules of the training course at their work place and during their work shift so they will have to be released from their clinical duty only 30 minutes at a time.
  Interventions: Other: longitudinal NRP training

INTERVENTIONS:
Other: Single-day NRP Training — NRP training course completed in one single day of 8 hours
  Arms: Single-day NRP training
Other: longitudinal NRP training — NRP training course completed over one year by attending nine 30-minute modules.
  Arms: Longitudinal one year NRP Training

SUMMARY:
The Neonatal Resuscitation Program (NRP) recommends providers renew their certification every 2 years. However, many Neonatal Intensive Care Units (NICUs) in Canada face challenges of significant budget cuts in training and a large number of caregivers to train with a high turnover rate. This situation makes it difficult for managers and nurse educators to ensure up-to-date certification and competence for all clinical staff. In addition, considering that only 0.1% of newborns will require cardiac massage and/or epinephrine, health care professionals' exposure to critical events is low to insure maintenance of expertise. Furthermore, it is shown that there is a significant decrease in knowledge among learners who have undergone specific training after only 3 months. This is worrisome considering that some nurses will not renew their certification if the course is not paid for by the employer, or if they are not released from clinical duties to attend. While keeping in mind the various required components of NRP training: book reading, online exam, performance stations, Integrated Skills Station Assessment (ISSA) and simulations, we would like to assess the educational and financial impact of a new educational strategy developed as to allow more nurses to be retrained thus ensuring maintenance of their neonatal resuscitation expertise.

ELIGIBILITY:
Inclusion Criteria:

* Newly recruited ( in the last 3 months) neonatal and delivery room registered nurses from level 2 and 3 perinatal centers

Exclusion Criteria:

* Registered nurses that have already completed a NRP training in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 1 year
  Integrated Skills Stations Assessment Score. The higher the score, the better the performance. Scores range from 0 to 100 %.

SECONDARY OUTCOMES:
Confidence and behavior | 1 year
  continuing professional development (CPD) reaction questionnaire (REACT). The higher the score, the better the outcome. Scores range from 12 to 82.
Cost-efficiency | 1 year
  Cost of each educational intervention (each arm).

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Cité de la santé de Laval, Laval, Quebec
  - University of Montreal Health Center, Montreal, Quebec
  - CHU Sainte-Justine, Dept Neonatology, Montreal, Quebec
  - CHUL, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
  - Jewish General Hospital, Montreal
  - Pierre-Legardeur, Repentigny

IPD SHARING:
Plan to Share IPD: No